CLINICAL TRIAL: NCT02987647
Title: Phase IV Pilot, Longitudinal, Prospective, Double-blind, Comparative to Assess the Perception of Efficacy, Safety and Tolerability of Three Non-hormonal Intravaginal Gels and Hormone Cream in Postmenopausal Women
Brief Title: Perception of Efficacy, Safety and Tolerability of Three Non-hormonal Intravaginal Gels and Hormone Cream
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Farmoquimica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HIDRAPILOTO
Record Dates: First submitted 2016-11-03; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Vaginal Dryness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Hidrafemme (Experimental): The arm in question will have 14 patients who use the Hidrafemme product, encoded as group A.
  Name: hidrafemme Dosage form: applicator Dosage: the applicator must be complete (full) Frequency: twice a week Duration: 28 days
  Interventions: Other: Hidrafemme
- Vagidrat (Active Comparator): The arm in question will have 14 patients who use the Vagidrat product, encoded as group B.
  Name: vagidrat Dosage form: applicator Dosage: the applicator must be complete (full) Frequency: twice a week Duration: 28 days
  Interventions: Other: Vagidrat
- Lubrinat (Active Comparator): The arm in question will have 14 patients who use the Lubrinat product, encoded as group C.
  Name: lubrinat Dosage form: applicator Dosage: the applicator must be complete (full) Frequency: twice a week Duration: 28 days
  Interventions: Other: Lubrinat
- Antrofi (Active Comparator): The arm in question will have 14 patients who use the Antrofi product, encoded as group D.
  Name: antrofi Dosage form: applicator Dosage: the applicator must be complete (full) Frequency: twice a week Duration: 28 days
  Interventions: Other: Antrofi

INTERVENTIONS:
Other: Hidrafemme — The complete treatment will have followed four weeks of duration and application of the product should take place twice a week.
  Arms: Hidrafemme
Other: Vagidrat — The complete treatment will have followed four weeks of duration and application of the product should take place twice a week.
  Arms: Vagidrat
Other: Lubrinat — The complete treatment will have followed four weeks of duration and application of the product should take place twice a week.
  Arms: Lubrinat
Other: Antrofi — The complete treatment will have followed four weeks of duration and application of the product should take place twice a week.
  Arms: Antrofi

SUMMARY:
To evaluate the perception of the effectiveness of Hidrafemme® gels, Vagidrat®, Lubrinat and Antrofi cream in improving vaginal moisture in postmenopausal women who are currently registered options most current and available in the market in order to assess the differences between them, subsequently conduct a clinical study larger.

DETAILED DESCRIPTION:
Before any procedure of the study, the researcher should have undertaken a detailed discussion on the Consent and Informed remedying any questions the patient may present. Then the principal investigator and the patient must sign all pages of the Consent and Informed (two-way), each one with a copy. Female patients aged above 40 years postmenopausal and who are diagnosed with vaginal dryness, will be invited to participate in this study. After the selection, through the inclusion and exclusion criteria, and signing the consent form Clarified, research participants will be evaluated by clinical examination (VHI), pH evaluation (using pH tape), questionnaire application IFSF and subjective evaluation of the patient. All the above procedures will be performed in own research center for the study team. The study in question has four (4) treatment groups with fourteen (14) patients each, totaling fifty-six (56) patients. The allocation of these patients will occur blind, parallel to the first group use the Hidrafemme, the second uses the Vagidrat, uses the third and fourth Lubrinat use the Antrofi. All groups conduct the use of those products, twice a week for four (4) consecutive weeks. After the addition, the research participant will receive the product under study and will be oriented as their dosage, correct application form and the records in the patient diary.

After the Visit 1 (initial) the research participant must return for another visit in person, Visit 2 (final), the research center, which will take place 28 calendar days after the date of Visit 1 (initial). During all the above visits, the participants research will be assessed by the principal investigator and will be conducted the subjective evaluation of the patient, VHI evaluation (attached), pH control and will fill the IFSF form (attached). At the final visit will be also evaluated the acceptability of the product and adherence to treatment through the patient diary. The adverse event occurrences will be evaluated during the final visit. If any research participant submit an adverse event, it will be accompanied by research center staff to its resolution. The variables related to the effectiveness of the product will be studied by VHI scale, which indicates the score of each item under study. The score should be evaluated for each variable. Daily application for registration throughout the period of four (4) weeks, and the product will be dispensed after the inclusion / randomization of the patient during the initial visit, sufficient to twenty-eight (28) days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 40 years.
* Healthy Women of post-menopausal (no period for more than one year).
* Women with vaginal dryness.
* Women with active sex lives of at least 1 sexual intercourse in the month.
* Women without a history of sensitivity.
* Understanding and signing the Consent and Informed.

Exclusion Criteria:

* Women in use of any intravaginal moisturizing gel, vaginal cream and / or spermicide.
* Women with a diagnosis or history of cancer.
* Women with disease or condition that, in the opinion of the gynecologist, could affect the study results.
* Women using hormone replacement therapy in the last 3 months.
* History or visible evidence of chronic skin disease or regional infections.
* History of hypersensitivity (allergy) to promestrieno.
* Women with genital herpes, vaginal infections or urinary tract infection.
* Pregnant women and nursing mothers.
* Allergy Personal history and hypersensitivity to any feminine hygiene product.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Categories VHI scale for intensity of vaginal moisture | 28 days
  The efficacy parameter: intensity of vaginal moisture; It will be measured by the VHI: 1 = no / inflamed surface; 2 = no / not inflamed surface; 3 = minimal, 4 = moderate, 5 = Normal. They will be described by mean and standard deviation or median and interquartile range, as well as minimum and maximum. If there is a normal distribution and equal variance will be held the Split-Plot ANOVA measures and where there are significant differences will be a post hoc Tukey and Dunnet. 95% confidence intervals for the mean difference will be calculated

SECONDARY OUTCOMES:
Score the increase in Sexual Function Index Women | 28 days
  The score index of female sexual function (SIFIs) will be described on a monthly basis by mean and standard deviation or median and interquartile range, as well as minimum and maximum. If there is a normal distribution and equal variance will be held the Split-Plot ANOVA test and if there are no significant differences will be performed post hoc Tukey and Dunnet as appropriate. 95% confidence intervals for the mean differences in each visit will be calculated.
pH vaginal | 28 days
  It will be measured by its own value, described on a monthly basis by mean and standard deviation or median and interquartile range, as well as minimum and maximum. If there is a normal distribution and equal variance will be held the Split-Plot ANOVA test and if there are no significant differences will be performed post hoc Tukey and Dunnet as appropriate. 95% confidence intervals for the mean differences in each visit will be calculated.
Acceptability of the product | 28 days
  The acceptability of the product will be assessed by the patient using a satisfaction scale: 1 = very satisfied, 2 = satisfied, 3 = makes no difference, 4 = dissatisfied and 5 = very dissatisfied And others.
Subjective patient evaluation | 28 days
  Patients will assess all visits the intensity of itching and stinging / burning of the vagina on a scale such as: 1 = Severe 2 = Moderate; 3 = mild; 4 = no For the variables: Fire / vaginal burning will be summed up at all visits, in terms of mean and sta or Kruskal-Wallis depending on if there is a normal distribution and equal variance.

CONTACTS AND LOCATIONS:
Overall Officials: Thales Braga, analist, Study Director — FQM

IPD SHARING:
Plan to Share IPD: No